CLINICAL TRIAL: NCT04303052
Title: Randomized-Controlled Non-Inferiority Study to Compare the Effectiveness of the Seldinger Over-the-Wire Technique and the Modified Seldinger Technique
Brief Title: Non-Inferiority Study to Compare the Effectiveness of the Seldinger Over-the-Wire Technique and the Modified Seldinger Technique
Acronym: Over-the-Wire
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jena University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5385-12/17
Record Dates: First submitted 2019-03-12; First posted 2020-03-10 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Effectiveness and Safety of the Seldinger Wire Technique Using a 145 cm Guidewire With the Modified Seldinger Technique Using a 70 cm Guidewire

STUDY DESIGN:
Intervention Model Description: Depending on randomization, the Power-PICC implantation occurs either with Seldinger over-the-wire technique or with Seldinger modified technique. All related substances, measures or procedures are performed according to the clinical routine.
Who Masked: Participant
Masking Description: On the intervention day, the patient is randomly assigned to one of the two study arms through envelope (145 cm vs 70 cm)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- over-the-wire technique with 145 cm guidewire (Active Comparator): Catheter tip placement using Seldinger over-the-wire technique with 145 cm guidewire
  Interventions: Device: Angiodynamic Bioflo Picc IR-KIT (145 cm guidewire) or
- modified technique with 70 cm guidewire (Active Comparator): Catheter tip placement using Seldinger modified technique with 70 cm guidewire
  Interventions: Device: Angiodynamic Bioflo Picc MST-KIT (70 cm guidewire)

INTERVENTIONS:
Device: Angiodynamic Bioflo Picc IR-KIT (145 cm guidewire) or — Before Power-PICC-line catheter implantation, the patients undergo an examination of the planned intervention site and ultrasound check, and analysis of the blood tests. An informed consent discussion and the patient's signature on the informed consent are obligatory. The length of the catheter and the optimal position of the catheter tip are verified by fluoroscopy. After catheter implantation, the tip location is verified by a final chest x-ray. The follow-up visit and the control of the puncture site until removal of the catheter are performed during hospitalization or subsequently by the treating family doctor.
  Arms: over-the-wire technique with 145 cm guidewire
Device: Angiodynamic Bioflo Picc MST-KIT (70 cm guidewire) — Before Power-PICC-line catheter implantation, the patients undergo an examination of the planned intervention site and ultrasound check, and analysis of the blood tests. An informed consent discussion and the patient's signature on the informed consent are obligatory. The length of the catheter and the optimal position of the catheter tip are verified by fluoroscopy. After catheter implantation, the tip location is verified by a final chest x-ray. The follow-up visit and the control of the puncture site until removal of the catheter are performed during hospitalization or subsequently by the treating family doctor.
  Arms: modified technique with 70 cm guidewire

SUMMARY:
Peripherally inserted central venous catheter lines (PICC-line) are successfully used since many years in patients who need long-term frequent IV therapy. The PICC placement is performed under fluoroscopy The study objective is to compare the effectiveness and safety of the Seldinger wire technique (over-the-wire) using a 145 cm guidewire with the modified Seldinger technique using a 70 cm guidewire.

DETAILED DESCRIPTION:
The referral of patients with indication to PICC-line implantation at the institute of diagnostic and interventional radiology occurs through different departments of the University Hospital Jena. The patients are registered for radiological treatment and checked again by a radiologist if a PICC-line implantation is indicated. If this is the case, the radiologist conducts an informed consent discussion with the patient about possible complications and risks during intervention and informs him also about a possible study participation. After signature of the written informed consent, the patient is included. He can, at any time, withdraw his consent. On the intervention day, the patient is randomly assigned to one of the two study arms through envelope (145 cm vs 70 cm). The intervention time is documented. After intervention, the patient is transferred back to the ward or sent home. The examination of the puncture site before discharge is performed by a ward physician or by the family doctor.

Within 2 weeks after PICC-line implantation, the treating physician is contacted and questioned about possible complications (catheter occlusion, haematoma, infection of the puncture site, arm vein thrombosis, pain, etc.), that are then thoroughly documented.

ELIGIBILITY:
Inclusion Criteria:

* female, male
* adults ≥ 18 years
* medical indication for Power-PICC-Line catheter implantation because of chemotherapy or parenertal nutrition
* in- and outpatients

Exclusion Criteria:

* age < 18 years
* systemic infection
* local infection of the interventional location
* known allergy to used material
* general contraindication of Power-PICC-Line catheter implantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2018-02-02 (Actual); Primary Completion 2019-08-28 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Implantation time | 24 hours
  Economy of time until beginning of treatment

SECONDARY OUTCOMES:
Placement accuracy of catheter tip compared to chest x-ray | 24 hours
  by final chest X-ray

CONTACTS AND LOCATIONS:
Overall Officials: Heike Habrecht, Dr., Principal Investigator — Institute of Diagnostic and Interventional Radiology
Locations (1):
- University Hospital Jena, Jena, Thuringia, Germany